CLINICAL TRIAL: NCT06417151
Title: Comprehensive Dietary Assessment of Children Aged 1 Year to 6 Years (5-72 Months) - a Cross-sectional, Nationwide Study: PITNUTS 2024
Brief Title: Polish Infants and Toddler Nutritional Study
Acronym: PITNUTS
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundacja Nutricia (Other)
Collaborators: Institute of Mother and Child, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 40/2024; RG 1/2023 (Other Grant/Funding Number: Fundacja Nutricia)
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Diet Habit; Dietary Habits; Diet, Healthy; Children; Child; Nutritional Deficiency; Nutritional Status; Macronutrients; Consumption; Dietary Assessment; Cross-sectional Study
Keywords: diet; habit; nutritional; children; cross-sectional study; macronutrients; child; dietary assessment; consumption
MeSH Terms: conditions — Feeding Behavior; Malnutrition; Habits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children between the ages of 5 months and 6 years of Polish nationality

SUMMARY:
A cross-sectional study representative of the Polish population of children aged 5 months to 6 years conducted in the cross-sectional study model, the main objective of which is to assess the nutritional value of the diet of children aged from 5 months to 6 years with regard to the basic macronutrients: protein (P), fat (F), carbohydrates (C). The study will include: dietary interviews, which will include the Food Frequency Questionnaire questionnaire (FFQ) and a 3-day food diary, as well as anthropometric measurements. The study will involve 1,000 children who will be selected by a random draw based on government database. The survey will be conducted by trained field interviewers - training will be provided by a dietician and an anthropologist. The study also included validation of the FFQ questionnaire.

DETAILED DESCRIPTION:
Background:

Correct nutrition is one of the most important factors for the optimal psychosomatic development of the child. Both short- and long-term observations emphasise the importance of nutritional factors in the childs development already in the foetal period and in the first two years of life (the idea of the first 1,000 days of life). Research shows that the components of the model of safe child nutrition, such as exclusive breastfeeding of the child in the first six months of life, breastfeeding and skilful expansion of the diet in the second six months of life and appropriate nutritional management in the post-natal and pre-school period form the basis for normal growth, the formation of healthy eating behaviour and also reduce the risk of diet-related diseases in adulthood. Parental awareness towards skilful dietary expansion and the introduction of foods with a favourable nutrient profile depends to a large extent on effective nutrition education (PITNUTS 2016). Data on infant and child nutrition in Poland are limited. The PITNUTS study, conducted in Poland in 2016 on a randomly selected sample (N=1059), found that the diet of infants and children aged 5-36 months deviated from the dietary recommendations. An analysis of the nutrient profile in the diets of postnatal children showed a varied energy value and a significantly higher protein supply in relation to population norms (Weker et al, 2017; Weker et al, 2019). A survey conducted during the COVID-19 pandemic by Horvath et al. also showed a discrepancy between mothers; nutritional knowledge and feeding practices of infants aged 4-12 months (Horvath et al, 2022). Inappropriate feeding practices translated into nutritional status, which was confirmed in a study conducted in Poland as part of the National Health Programme 2016-2020 (Kułaga ed. 2021). On the other hand, in a nationwide study conducted in 2017-2020 among pre-school and school children, abnormal body weight was found in more than 30% of respondents (PAN 2023). Observational studies conducted worldwide have confirmed the short- and long-term effects of nutrition on the nutritional status of infants and young children. A beneficial effect of diets including fortified foods on reducing the risk of deficiencies of nutrients such as iron, vitamin D and calcium and the energy balance of the diet has also been found (Lioret et al 2015, Schroeder et al 2015, Ahluwalia et al 2016, Hammer et al 2016, Akkermans et al 2017, McCarthy 2017, Finn et al 2017, Csölle Iet al 2022).

In recent years, updated and revised dietary recommendations for the paediatric population, for three age groups, have been issued, based on the latest reports and international recommendations (Fewtrell et al 2017, Hojsak et al 2018, Fidler et al 2017, Dereń et al 2019).

Updated Guidelines of nutrition for healthy infants - Position statement of the Polish Society of Gastroenterology, Hepatology and Child Nutrition, in line with current ESPGHAN guidelines, the Position statement of the Committee on Human Nutrition Science of the Polish Academy of Sciences on the principles of nutrition for children aged 1-3 years and the Position statement of the Committee on Human Nutrition Science of the Polish Academy of Sciences on the principles of nutrition for pre-school (4-6 years) and early school age children (7-9 years) were developed. Changes to the guidelines included, among others, the introduction of allergenic foods, the serving of plant-based beverages and fruit juices (in the first year of life), and the updating of safe nutrition models in relation to food rations (in the 1-3 years and 4-9 years groups) (Szajewska H. et al, 2021, PAN 2022, PAN 2023).

Understanding current practices and challenges in infant and child nutrition will allow better tailoring of nutrition education interventions targeting parents and children. The aim of this study is to assess the diet and nutritional status of infants and children aged 5-72 months, the consistency of feeding practices with current recommendations and to compare with the results of the previous PITNUTS survey conducted in 2016.

On this basis, investigators hypothesise that children aged 5 months to 6 years are not fed according to the principles of proper nutrition (Szajewska et al. 2021 , Weker et al. 2022 , Weker et al.2023 , Jarosz M. et al. 2020 ], and their nutritional status assessed on the basis of anthropometric measurements deviates from the norms based on the WHO centile grids for children 0-5 and for children ≥3 years of age OLA-OLAF (Kułaga 2015).

Objectives:

The main objective of the study is to assess the nutritional value of the diet of children aged 5 months to 6 years with regard to the main macronutrients: protein (B), fat (T), carbohydrates (C). In addition, specific objectives were also identified:

* to assess the nutritional value of the diet in terms of other nutrients: animal protein, vegetable protein, digestible carbohydrates, dietary fibre, lactose, sucrose, starch, polyunsaturated fatty acids (PUFA), monounsaturated fatty acids (MUFA), saturated fatty acids (SFA), vitamins, minerals
* assessment of population risk of deficiencies based on nutrient intakes (cut-off point method [Estimated Average Requirement (EAR)/Adequate Intake (AI)], with particular reference to vitamin D, LCPUFA and protein
* assessment of nutritional status based on Z-score BMI, i.e. body mass index related to age and sex

Study Population:

The study will include healthy children aged 5 months to 6 years.

Sample sizes were determined in two ways:

First was ensuring that the results of the study can be generalized to the populations of children aged 5-12 months, 13-36 months and 37-72 months with a 95% confidence interval, and that the maximum assumed error (difference between the population parameter and the sample statistic) will not exceed 6%. The sample will be selected in such a way as to ensure both representativeness for the whole population (infants and children from the whole country at a specific age: 5 months - 6 years). The study will include all drawn children whose parents agree to participate in the study (informed consent form, parents/guardians of children drawn for the study will be offered a quota voucher to be used at a selected retail chain). The draw will be carried out in strata taking into account the age of the child and the type of municipality, and within a stratum, the draw of a specific bundle (municipality) will be carried out with probability proportional to the number of children aged up to six years old in the municipality (based on CSO data - Census 2021). As a result, also the number of bundles per province within the stratum will be roughly proportional to the number of children in the province and the type of municipality. The sample will comprise 300 infants aged 5-12 months, 400 children aged 13-36 months and 300 children aged 37-72 months. Infants up to the age of one year will be further stratified (5-6, 7-9 and 10-12 months with 100 infants each), children aged 13-36 months will be stratified by year: 13- 24 and 25-36 months (200 babies each), and children over 36 months into annual strata of 100 babies each. This scheme ignores the not-quite-uniform distribution of births across months and years, but taking it into account would be extremely difficult, as such detailed population data, even if it were possible to obtain in real time, loses relevance very quickly. The simplification adopted will have minimal impact on the quality of the sample, but will allow a minimum sample size of 100 interviews to be maintained for the narrowest ranges. Children will be selected on the assumption that they will be aged 4, 6, 9, 12, 24, 36, 48 and 60 months respectively on the day of the survey. The need to complete the survey in a short period of time due to sample obsolescence (the age of the children had to be within the assumed ranges) necessitates drawing an appropriately paired sample and providing an adequate reserve sample in case the child/carer did not agree to participate in the survey or was unavailable on the survey date. The municipality was used as the primary sampling unit. For operational reasons, two parallel representative samples of the original sampling units (municipalities) of 100 units each (sample A and sample B) will be drawn. In municipalities drawn into the first group (sample A), one interview each will be conducted with parents/carers of children from age cohorts 1a, 1c, 2a, 2b, 3b (subgroup designations as in the Table below). In municipalities from the second group (sample B) - one interview each with parents/carers of children from subgroups: 1b, 2a, 2b, 3a, 3c. This will yield as many interviews per age cohort as below:

1. Infants (n=300) 1a. Infants 5-6 months (n=100) 1b. Infants 7-9 months (n=100) 1c. Infants 10-12 months (n=100)
2. Children 13-36 months (n=400) 2a. Children 13-24 months (n=200) 2b. Children 25-36 months (n=200)
3. Children 37-72 months (n=300) 3a. Children 37-48 months (n=100) 3b. Children 49-60 months (n=100) 3c. Children 61-72 months (n=100)

In addition to ensuring representativeness, abundance was counted for the primary endpoint. For this purpose, P, F, C intake data from PITNUTS 2016 were used (mean and SD) for children 5-6 months, as this age group had the greatest variability in macronutrient intake. An acceptable error of 15% in the estimation of the mean value was assumed; the formulae for the quantitative data (mean and SD) were applied in the design of the descriptive studies. The results of these calculations indicated a minimum sample N calculated for the intake of P: 97; F: 91; C: 94 individuals. Therefore, the assumed sample size of 100 children aged 5-6 months is sufficient with an acceptable 15% error in the estimation of the mean value in this age group. On this a priori basis, similar counts were used for the other age groups, i.e. 100 or 200 individuals each. From the intake data obtained in PITNUTS 2016 and the a priori counts (100 or 200 individuals each), it was concluded that such counts in the age groups 7-9 mo, 10-12 mo and 5-12 mo would allow an estimate of the mean intake of P, F, C with an acceptable error in the range of 5-10%. After the fact, the power of the test for intake will be calculated from the intake data obtained in PITNUTS 2024 (to determine the power of inference in the main study) for the realised counts:

* P, F, C in the age groups 13-36 mo, 37-72 mo.
* other nutrients in all age groups
* percentage of people at risk of deficiency

In summary, the numbers of children aged 5-72 months in each age range will be:

* 5-12 months [1 year of age] (N=300, of which: 5-6 months =100, 7-9 months =100, 10-12 months =100)
* 13-36 months [2, 3 years of age] (N=400, of which: 13-24 months =200, 25-36 months =200)
* 37-72 months [4, 5, 6 years of age] (N=300, of which 37-48 months =100, 49-60 months =100, 61-72 months =100)

Research tools and methods:

The survey will be carried out by field interviewers who will have received prior training in nutrition interviewing and anthropometric measurements. The training will be provided by a dietician and an anthropologist.

The parent (legal guardian), together with the interviewer will fill in a survey questionnaire with the inclusion of a food frequency questionnaire (FFQ) computer-assisted personal interview (CAPI), aimed at a qualitative assessment of the diet, including the identification of eating patterns. The survey will also collect socio-demographic characteristics/family/environmental conditions.

A quantitative assessment of diet, including the nutritional value of diets will be assessed by recording food intake from 3 consecutive days, including one weekend day [a diet diary completed by the parent/legal guardian themselves] in an online format. The data will be entered into the Diet 6 program where the nutritional value of the diets from the individual diaries will be calculated. During the completion of the FFQ form, the interviewer will explain in detail how to complete the food diaries.

Anthropometric measurements will be taken using certified medical scales, growth meter and measurement pad. The measurements will be carried out by pre-trained interviewers who will also have detailed instructions on how to carry out the anthropometric measurements (prepared earlier by an anthropologist):

* for the 5-24 months group, measurements will be carried out in the supine position using the SECA 834 balance and the SECA 417 measuring pad
* for the group of 25 months to 6 years of age, measurements will be carried out in the standing position using the SECA 878 and the stadiometer SECA 217.

The results obtained will be entered by the interviewer in the anthropometric measurement record sheet.

Validation of the FFQ questionnaires:

Validation of the FFQ questionnaires will be carried out as part of the study. It is planned to use the FFQ questionnaire for groups: 5-12 mo. 13-36 mo., 37-72 mo. For all 3 groups, validation will be carried out by determining their internal FFQ concordance (reproducibility) on the following numbers:

- 5-12 mo. - 100 subjects; 13-36 mo. - 100 subjects; 37-72 mo. - 100 individuals. FFQ will be completed and administered by the same interviewer during the dietary interview twice, 14 days apart.

Statistical analysis plan:

1. Characterization of groups based on socio-demographic data: descriptive statistics, analysis of variable distributions, frequencies of socio-demographic characteristics
2. evaluation of the diet of the groups:

   a. Qualitative type data on feeding habits: structure indicators on number of feedings, introduction of complementary foods in the following months of infants; life, sweetening/salting of food, number of meals per day b. Qualitative type data collected by the food frequency method (from FFQ questionnaires): structure indicators for the frequency of consumption categories of the different food groups c. Data of quantitative type from the food record method (nutritional value of the diet of 3 days): - descriptive statistics, analysis of variable distributions, structure indicators for population risk of inadequate nutrient intake (i.e. determination of percentage of children): i. group average requirement standard (EAR) or below adequate intake standard (AI), e.g. for protein (EAR), ii. WHO recommended intake, e.g. for sucrose ≥10% of Energy, Cut-off points (EAR, AI, sucrose/added sugars ≥10%E) will be determined based on the Nutrition Standards for the Polish Population (2020) and WHO 2015 recommendations.

   d. Significance of difference tests to compare children of different age groups: comparison of population structure indicators of inadequate dietary risk, e. Significance of difference tests to compare children of the same age group with different degrees of fit to each identified DP (upper tercile vs lower tercile, upper tercile vs middle tercile): comparison of structure indicators on eating behavior, comparison of daily frequency of food intake, comparison of nutritional value of the diet, comparison of predefined dietary patterns (diet quality indicators)
3. assess the nutritional status of groups of children:

   1. Quantitative data (body weight, length/height, weight-to-length/height index, z-score weight-to-length/height, z-score-BMI): descriptive statistics, analysis of variable distributions
   2. Qualitative data: indices of the structure of the prevalence of nutritional status disorders according to WHO centile grids for children 0-5, OLA-OLAF for children ≥3 years of age (for children aged 0-35 months z-score weight-to-length/height categories or z-score BMI: (1) normal nutritional status ≥-2 SD to +1 SD; (2)possible risk of overweight 1 SD to 2 SD; (3) overweight 2 SD to 3 SD; (4) obesity (5) weight-to-length/height deficiency 2 SD to -3 SD; (6) significant weight-to-length/height deficiency -3 SD; for children ≥3 years of age, underweight, overweight and obesity categories as defined by OLA-OLAF grids based on z-score BMI
4. evaluation of the relationship between diet and nutritional status of children, taking into account the influence of associated variables (family-environmental determinants):

   1. tests of significance of differences to compare children with different nutritional status grouped according to the categories listed in the section Assessment of the nutritional status of groups of children: comparison of structure indicators on eating behavior, comparison of daily frequency of food intake, comparison of nutritional value of the diet, comparison of predefined dietary patterns (diet quality indicators), comparison of structure indicators of the incidence of population risk of inadequate intake;
   2. Significance of difference tests to compare children with different degrees of fit to predefined dietary patterns and fit to data-driven dietary patterns: comparison of structure indicators of the prevalence of nutritional status disorders according to WHO centile grids for children 0-5, OLA-OLAF for children ≥3 years of age (listed in the section ;Assessment of nutritional status of groups of children), comparison of structure indicators of the prevalence of population risk of inadequate intake (EAR/AI or recommended intake);
   3. Logistic regression analysis for modelling: population risk of inadequate nutrient intake (EAR/AI or recommended intake) according to socio-demographic characteristics of children/families, BMI of parents/guardians, nutritional knowledge of parents/guardians; chance of good dietary adjustment (upper tercile) depending on socio-demographic characteristics of children/family, BMI of parents/guardians, nutritional knowledge of parents/guardians; chance of good diet quality (upper tercile of healthy diet index) depending on socio-demographic characteristics of children/family, BMI of parents/guardians, nutritional knowledge of parents/guardians; the chance of poor diet quality (upper tercile of the unhealthy diet index) depending on socio-demographic characteristics of children/family, BMI of parents/guardians, nutritional knowledge of parents/guardians; the risk (with adjustment for socio-demographic characteristics of children/family, BMI of parents/guardians, nutritional knowledge of parents/guardians) of the occurrence of nutritional disorders (listed in the section ;Assessment of nutritional status of groups of children) depending on good adjustment to the dietary pattern (upper tercile)

ELIGIBILITY:
Inclusion Criteria:

* healthy children aged 5 months to 72 months born at term
* polish nationality

Exclusion Criteria:

* Presence of chronic diseases affecting nutritional status (metabolic diseases - e.g. diabetes, phenylketonuria, cystic fibrosis; diseases of the digestive system - e.g. coeliac disease, Crohn's disease; kidney disease, liver disease or other disorders affecting the absorption of nutrients)
* Use of elimination diets for medical reasons (e.g. food allergy)
* Developmental disorders that may affect nutrition (e.g. genetic diseases, prematurity)
* Acute infectious disease or other illness requiring hospital treatment within 3 months prior to the start of the study
* Condition after a prolonged hospital stay (>10 days) within 6 months prior to the study
* Surgical procedures performed in the last 3 months that could affect nutritional status

Ages: 5 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It will be children randomly selected from different socio-economic backgrounds. The sample will be drawn on the basis of PESEL numbers. The children surveyed will come from the whole area of Poland with territorial representativeness. The respondents in the survey will be parents or legal guardians of the drawn children. The division into age groups is based on the key stages of a child's development, i.e. up to 1 year of age (n=300), 1-3 years of age (n=400), after 3 years of age and up to 6 years of age (n=300).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Macronutrient intake | three-day consumption
  Nutritional value of the diet in terms of macronutrients: protein, fat, carbohydrates

SECONDARY OUTCOMES:
Other nutrients intake | three-day consumption
  Nutritional value of the diet in terms of other nutrients: animal protein, vegetable protein, digestible carbohydrates, dietary fibre, lactose, sucrose, starch, polyunsaturated fatty acids (PUFA), monounsaturated fatty acids (MUFA), saturated fatty acids (SFA), vitamins, minerals (as well as in terms to primary nutrients: protein, fat, carbohydrates) will be calculated (per person/day) using the computer program (DIETA 6, National Food and Nutrition Institute, Warsaw) including Polish food composition tables. To collect dietary data 3-day estimated food record (FR) will be used.
Population risk of nutritional deficiencies | the last 14 days of the FFQ
  Based on nutrient intake cut-off point method [Estimated Average Requirement (EAR)/Adequate Intake (AI)] with a focus on vitamin D, Long-Chain Polyunsaturated Fatty Acids (LCPUFA) and protein
Nutritional status | At the time of the dietary interview
  Assessment of nutritional status based on Z-score BMI, or body mass index related to age and sex

OTHER OUTCOMES:
Dietary regime | the last 14 days of the FFQ
  Number of meals and snacking
Frequency of food consumption | the last 14 days of the FFQ
  Frequency of food consumption based on data from the FFQ
Dietary Patterns | the last 14 days of the FFQ
  Dietary patterns identified by two methods: predefined (diet quality indicators) and data-based (principal component factor analysis)
Dietary supplements | the last 14 days of the FFQ and three-day consumption from food diaries
  use of dietary supplements in children based on FFQ and food diaries
Nutritional Knowledge | the last 14 days of the FFQ
  level of declared nutritional knowledge of parents from questionairre

CONTACTS AND LOCATIONS:
Locations (1):
- Mothers and Child Institute, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weker H, Brudnicka E, Baranska M, Rowicka G, Strucinska M, Wiech M, Dylag H, Klemarczyk W, Socha P, Mazur J. Dietary Patterns of Children Aged 1-3 Years in Poland in Two Population Studies. Ann Nutr Metab. 2019;75(1):66-76. doi: 10.1159/000501422. Epub 2019 Jul 2. PMID 31266006
- [Background] Weker H, Baranska M, Riahi A, Strucinska M, Wiech M, Rowicka G, Dylag H, Klemarczyk W, Bzikowska A, Socha P. Nutrition of infants and young children in Poland - Pitnuts 2016. Dev Period Med. 2017;21(1):13-28. doi: 10.34763/devperiodmed.20172101.1328. PMID 28551688
- [Background] Schroeder N, Rushovich B, Bartlett E, Sharma S, Gittelsohn J, Caballero B. Early Obesity Prevention: A Randomized Trial of a Practice-Based Intervention in 0-24-Month Infants. J Obes. 2015;2015:795859. doi: 10.1155/2015/795859. Epub 2015 May 11. PMID 26078877
- [Background] McCarthy EK, Ni Chaoimh C, Hourihane JO, Kenny LC, Irvine AD, Murray DM, Kiely M. Iron intakes and status of 2-year-old children in the Cork BASELINE Birth Cohort Study. Matern Child Nutr. 2017 Jul;13(3):e12320. doi: 10.1111/mcn.12320. Epub 2016 Aug 9. PMID 27501864
- [Background] Lioret S, Betoko A, Forhan A, Charles MA, Heude B, de Lauzon-Guillain B; EDEN Mother-Child Cohort Study Group. Dietary patterns track from infancy to preschool age: cross-sectional and longitudinal perspectives. J Nutr. 2015 Apr;145(4):775-82. doi: 10.3945/jn.114.201988. Epub 2015 Jan 28. PMID 25833780
- [Background] Hojsak I, Bronsky J, Campoy C, Domellof M, Embleton N, Fidler Mis N, Hulst J, Indrio F, Lapillonne A, Molgaard C, Vora R, Fewtrell M; ESPGHAN Committee on Nutrition. Young Child Formula: A Position Paper by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):177-185. doi: 10.1097/MPG.0000000000001821. PMID 29095351
- [Background] Hamner HC, Perrine CG, Scanlon KS. Usual Intake of Key Minerals among Children in the Second Year of Life, NHANES 2003-2012. Nutrients. 2016 Jul 30;8(8):468. doi: 10.3390/nu8080468. PMID 27483313
- [Background] Finn K, Callen C, Bhatia J, Reidy K, Bechard LJ, Carvalho R. Importance of Dietary Sources of Iron in Infants and Toddlers: Lessons from the FITS Study. Nutrients. 2017 Jul 11;9(7):733. doi: 10.3390/nu9070733. PMID 28696361
- [Background] Fidler Mis N, Braegger C, Bronsky J, Campoy C, Domellof M, Embleton ND, Hojsak I, Hulst J, Indrio F, Lapillonne A, Mihatsch W, Molgaard C, Vora R, Fewtrell M; ESPGHAN Committee on Nutrition:. Sugar in Infants, Children and Adolescents: A Position Paper of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2017 Dec;65(6):681-696. doi: 10.1097/MPG.0000000000001733. PMID 28922262
- [Background] Lapillonne A, Bronsky J, Campoy C, Embleton N, Fewtrell M, Fidler Mis N, Gerasimidis K, Hojsak I, Hulst J, Indrio F, Molgaard C, Moltu SJ, Verduci E, Domellof M; ESPGHAN Committee on Nutrition. Feeding the Late and Moderately Preterm Infant: A Position Paper of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2019 Aug;69(2):259-270. doi: 10.1097/MPG.0000000000002397. PMID 31095091
- [Background] Deren K, Weghuber D, Caroli M, Koletzko B, Thivel D, Frelut ML, Socha P, Grossman Z, Hadjipanayis A, Wyszynska J, Mazur A. Consumption of Sugar-Sweetened Beverages in Paediatric Age: A Position Paper of the European Academy of Paediatrics and the European Childhood Obesity Group. Ann Nutr Metab. 2019;74(4):296-302. doi: 10.1159/000499828. Epub 2019 Apr 23. PMID 31013493
- [Background] Csolle I, Felso R, Szabo E, Metzendorf MI, Schwingshackl L, Ferenci T, Lohner S. Health outcomes associated with micronutrient-fortified complementary foods in infants and young children aged 6-23 months: a systematic review and meta-analysis. Lancet Child Adolesc Health. 2022 Aug;6(8):533-544. doi: 10.1016/S2352-4642(22)00147-X. Epub 2022 Jun 24. PMID 35753314
- [Background] Akkermans MD, Eussen SR, van der Horst-Graat JM, van Elburg RM, van Goudoever JB, Brus F. A micronutrient-fortified young-child formula improves the iron and vitamin D status of healthy young European children: a randomized, double-blind controlled trial. Am J Clin Nutr. 2017 Feb;105(2):391-399. doi: 10.3945/ajcn.116.136143. Epub 2017 Jan 4. PMID 28052885
- [Background] Ahluwalia N, Herrick KA, Rossen LM, Rhodes D, Kit B, Moshfegh A, Dodd KW. Usual nutrient intakes of US infants and toddlers generally meet or exceed Dietary Reference Intakes: findings from NHANES 2009-2012. Am J Clin Nutr. 2016 Oct;104(4):1167-1174. doi: 10.3945/ajcn.116.137752. Epub 2016 Sep 14. PMID 27629049
- [Derived] Sawicki M, Kowalkowska J, Kulaga Z, Socha P, Swiader-Lesniak A, Swiecicka-Ambroziak A, Szajewska H, Wadolowska L, Weker H. Assessment of dietary practices and nutritional status of children aged 5 to 72 months: study protocol of a nationwide Polish cross-sectional study (PITNUTS 2024). BMJ Open. 2025 Nov 19;15(11):e100921. doi: 10.1136/bmjopen-2025-100921. PMID 41263840